CLINICAL TRIAL: NCT04103398
Title: TRansarterial ChEmoembolization Plus SorAfenib Versus Transarterial Chemoembolization Alone for Recurrent Intermediate Hepatocellular Carcinoma: A Phase 3, Open Label, Multicenter, Randomized Controlled Trial
Brief Title: TACE Plus Sorafenib Versus TACE Alone for Recurrent Intermediate Hepatocellular Carcinoma
Acronym: TREAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, The vice president, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190921
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma; Sorafenib; Transarterial Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transarterial chemoembolization combined with sorafenib (Experimental): The initial dose of sorafenib is 400mg BID and the drug therapy will last till outcome events happen or the trial ends. TACE will start one day following oral sorafenib. Either conventional TACE (cTACE) or drug-eluting beads TACE (dTACE) is optional. TACE will be performed via injecting chemotherapy drugs (doxorubicin 50mg for cTACE or 75mg for dTACE) and embolizing agents (gelatin sponge for cTACE or microsphere for dTACE) into blood vessels that help tumor grow.
  Interventions: Combination Product: TACE+sorafenib
- Transarterial chemoembolization alone (Active Comparator): Either conventional TACE (cTACE) or drug-eluting beads TACE (dTACE) is optional. TACE will be performed via injecting chemotherapy drugs (oxaliplatin 200mg, raltitrexed 4mg, epirubicin 20mg in cTACE or 70mg in dTACE) and embolizing agents (gelatin sponge for cTACE or microsphere for dTACE) into blood vessels that help tumor grow.
  Interventions: Procedure: TACE

INTERVENTIONS:
Combination Product: TACE+sorafenib — The initial dose of sorafenib is 400mg BID and the drug therapy will last till outcome events happen or the trial ends. TACE will start one day following oral sorafenib. Either conventional TACE (cTACE) or drug-eluting beads TACE (dTACE) is optional. TACE will be performed via injecting chemotherapy drugs (doxorubicin 50mg for cTACE or 75mg for dTACE) and embolizing agents (gelatin sponge for cTACE or microsphere for dTACE) into blood vessels that help tumor grow.
  Arms: Transarterial chemoembolization combined with sorafenib
Procedure: TACE — Either conventional TACE (cTACE) or drug-eluting beads TACE (dTACE) is optional. TACE will be performed via injecting chemotherapy drugs (doxorubicin 50mg for cTACE or 75mg for dTACE) and embolizing agents (gelatin sponge for cTACE or microsphere for dTACE) into blood vessels that help tumor grow.
  Arms: Transarterial chemoembolization alone

SUMMARY:
The study is a multicenter phase III randomized trial. The purpose is to investigate both the efficacy and safety of transarterial chemoembolization (TACE) plus sorafenib versus TACE alone for recurrent intermediate hepatocellular carcinoma patients.

DETAILED DESCRIPTION:
The trial will recruit 162 patients with recurrent intermediate HCC, and they will be randomized (1:1) into two groups (TACE+sorafenib group, TACE group). Patients in TACE+sorafenib group will receive TACE one day following oral sorafenib (initial dose: 400mg BID). Patients in the TACE group will receive TACE alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years;
2. Diagnosed as HCC based on the American Association for the Study of Liver Diseases 2018 Guideline on Liver Cancer Diagnosis;
3. Initial tumor recurrence following curative surgical resection (R0 hepatectomy) (two to three lesions with at least one lesion >3 cm in diameter or more than three lesions of any diameter). Tumor burden ≤ 50% and no distant metastasis and macroscopic vascular invasion;
4. Histologically confirmed microvascular invasion in the specimen slices of surgically removed primary tumor;
5. Eastern Cooperative Oncology Group scoring 0-1;
6. Child-Pugh A class;
7. At least 3 months of life expectancy;
8. Adequate hematologic, hepatic and renal function: absolute neutrophil count ≥ 1.5x10^9/L, platelet ≥ 60 x10^9/L, Hb ≥ 90g/L, albumin ≥ 30g/L, total bilirubin ≤ 1.5 x upper limit of normal (ULN) , ALT < 5×ULN, AST < 5×ULN, alkaline phosphatase < 4×ULN, extended prothrombin time not exceeding 6s of ULN, creatine<1.5×ULN.

Exclusion Criteria:

1. Have lesions which are diffuse or can not be evaluated via imaging. Tumor burden>50%;
2. Have a history of hepatic encephalopathy, refractory ascites, severe esophageal and gastric varices or variceal bleeding and obstructive jaundice;
3. Have contraindications for TACE;
4. Have metastasis in central nervous system;
5. Allergic to intravenous contrast agents;
6. Pregnant or breastfeeding women, or expecting to conceive or father children within two years;
7. Infection of HIV, known syphilis requiring treatment;
8. Have a known history of prior invasive malignancies within 5 years before enrolment;
9. Patients with allotransplantation;
10. Severe dysfunction involving heart, kidney or other organs;
11. Severe active clinical infection which is over grade 2 based on NCI-CTC version 4;
12. Patients with mental disorders which may impact informed consent;
13. Unable to orally take drugs;
14. Participating other clinical drug trials 12 months before enrolment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  Defined as the time from randomization until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  Defined as the time from randomization until disease progression or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.
Time To Progression | 2 years
  Defined as the time from randomization until disease progression.
Objective Response Rate | 2 years
  The ratio of patients with complete response or partial response among all patients.
Disease Control Rate | 2 years
  The ratio of patients with complete response, partial response or stable disease among all patients.
Adverse Events | 2 years
  Grade 3 or severer hematological or non-hematological adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 4).
Scoring of Quality of Life | 2 years
  Using the third edition of European Organisation for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan W, Zhu B, Chen S, Wu Y, Zhao X, Qiao L, Huang Z, Tang R, Chen J, Lau WY, Chen M, Li J, Kuang M, Peng Z. Survival in Patients With Recurrent Intermediate-Stage Hepatocellular Carcinoma: Sorafenib Plus TACE vs TACE Alone Randomized Clinical Trial. JAMA Oncol. 2024 Aug 1;10(8):1047-1054. doi: 10.1001/jamaoncol.2024.1831. PMID 38900435